CLINICAL TRIAL: NCT00585962
Title: A Phase II Study Using Proton Beam Radiation Therapy for Early Stage Adenocarcinoma of the Prostate
Brief Title: Proton Beam Radiation Therapy for Early Stage Adenocarcinoma of the Prostate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American College of Radiology Imaging Network (Network)
Responsible Party: Principal Investigator, Anthony Laurence Zietman, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-064
Record Dates: First submitted 2007-12-27; First posted 2008-01-04 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer
Keywords: proton beam radiation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: Proton Beam Radiation — Once a day, 5 days a week (Monday-Friday), for 8 weeks.

SUMMARY:
The primary purpose of this study is to determine if high doses of radiation using proton beam can be given safely with low and acceptable side effects. This study will also gather data to determine the ability of the proton beam to eradicate prostate cancer. Proton beam radiation is a very accurate kind of treatment that has been shown to affect less normal tissue than a regular radiation beam.

DETAILED DESCRIPTION:
* Radiation therapy to the pelvis and prostate will be given once a day, 5 days a week (Monday-Friday), for 8 weeks. Each treatment takes about 10-20 minutes.
* Participants will be seen once a week for the entire 8 weeks by their study doctor to monitor and record any side effects. At the end of radiation therapy, participants will have a history and physical examination. Follow-up visits with the study doctor will be done at weeks 13 and 26 and then every 6 months for 3 years, then annually to year five.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously treated adenocarcinoma of the stages T1c-T2b and Gleason of equal to or greater than 5.
* PSA values of equal to or less than 15 ng/ml must be demonstrated within two months prior to study entry and greater than 3 weeks after prostate biopsy.
* Zubrod status 0-1.
* No evidence of distant metastasis.
* No evidence of other cancer. Prior malignancy does not exclude the patient if disease free for greater than five years.

Exclusion Criteria:

* Clinical stages T2c or above.
* PSA greater than 15.
* Any patient with T1c disease, a PSA less than or equal to 4 and Gleason sum less than 6.
* Evidence of lymph node involvement if lymph node sampling performed.
* Previous prostate surgery to include: simple prostatectomy, TURP, hyperthermia and cryosurgery.
* Previous prostate radiation.
* Prior hormonal therapy.
* History of inflammatory bowel disease even if currently inactive or controlled on medication.
* Prior systemic chemotherapy.
* History of proximal urethral stricture requiring dilatation.
* Current and continuing anticoagulation with Coumadin or equivalent.
* Major medical or psychiatric illness

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2004-02; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
To assess the late morbidity of 82 GY delivered to the prostate and surrounding tissues using proton beam radiation | 3 years

SECONDARY OUTCOMES:
To assess the acute morbidity following protocol treatment and to determine the ability of this treatment to control cancer. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Zietman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States